CLINICAL TRIAL: NCT00852280
Title: Effects of Pulsed-Dyed Laser on Scar Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, John Kevin Bailey, J. Kevin Bailey, MD Staff Surgeon, Shriners Hospitals for Children
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 08-6-24-1
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2010-07

CONDITIONS: Scars
Keywords: scars; late effect of burn; burn; pulsed-dye laser
MeSH Terms: conditions — Cicatrix; Burns | interventions — Lasers, Dye

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Treatment of 1/2 of skin graft with pulsed-dye laser — Pulsed-dye laser will be applied to 1/2 of the seam of the skin graft, using a 10mm spot size, and sufficient pulse-width and fluency to induce purpura.

SUMMARY:
The purpose of this study is to identify changes in color, thickness, and stiffness, of scars from skin grafting after burns when treated with a pulsed-dyed laser.

DETAILED DESCRIPTION:
Pulsed-dyed lasers have been used in the past to treat scars from minor surgery as well as burns. The laser has been used at different times, close to injury or late after injury. Success or failure of the laser has been judged by subjective observer scales.

In this study we will treat the seams of 1/2 of a skin graft with a pulsed-dyed laser, beginning about one month after surgery. We will use objective measures of color (redness on digital pictures), scar volume(via laser scanning), and elasticity(measured by BTC-2000) as well as subjective assessment by an independent observer and the patient.

ELIGIBILITY:
Inclusion Criteria:

* > 9 years old
* not pregnant
* new skin graft to extremity
* able to follow simple instructions

Exclusion Criteria:

* age less than 9 years
* pregnancy
* any behavior pattern that would lead to conclusion that patient may not reliably follow simple instructions

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Amount of redness of scar | 4 to 12 months after skin grafting

SECONDARY OUTCOMES:
Scar height | 4-12 months after skin grafting
Scar stiffness | 4-12 months after skin grafting
Patient's assessment of cosmetic outcome | 4-12months after skin grafting
Clinical improvement of appearance of scars assessed by subjective scale | 4-12 months after skin grafting

CONTACTS AND LOCATIONS:
Overall Officials: John K Bailey, MD, Principal Investigator — Shriners Hosptials for Children
Locations (1):
- Shriners Hospitals for Children, Cincinnati, Cincinnati, Ohio, United States